CLINICAL TRIAL: NCT05623046
Title: Building Emotional Self-Awareness Teletherapy (BEST): a Tool to Optimize Psychological Health Outcomes for Persons with Traumatic Brain Injury
Brief Title: Building Emotional Self-Awareness Teletherapy (BEST)
Acronym: BEST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Intrepid Center of Excellence (U.S. Federal Agency); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Flora Hammond, Chair of Department of Physical Medicine and Rehabilitation, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15355; W81XWH-22-2-0064 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2022-11-14; First posted 2022-11-21 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Concussion, Mild; Concussion, Brain; Concussion, Severe; Concussion, Intermediate; Concussion; Syndrome; Concussion Injury of Cerebrum; Concussion with Brief Loss of Consciousness; Alexithymia
Keywords: Alexithymia; Brain Injury; Concussion; Emotion Dysregulation; Affect; Resilience; Military; Service Members; Mood; Teletherapy
MeSH Terms: conditions — Brain Concussion; Syndrome; Affective Symptoms; Brain Injuries | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): 8 one-on-one teletherapy training sessions to enhance emotional skills. Teletherapy sessions will last approximately 60-90 minutes.
  Interventions: Behavioral: Treatment

INTERVENTIONS:
Behavioral: Treatment — 8 one-on-one teletherapy training sessions to enhance emotional skills. Teletherapy sessions will last approximately 60-90 minutes

SUMMARY:
To examine the feasibility, acceptability, and preliminary efficacy of a remotely delivered intervention for civilians and service members with mild traumatic brain injury (mTBI) who have difficulty recognizing and regulating their emotions. Post-treatment outcomes of interest include emotional self-awareness and regulation, resiliency, and affective symptoms.

DETAILED DESCRIPTION:
This Phase I proof of principle pilot study of the Building Emotional Self-awareness Teletherapy (BEST) intervention will use a quasi-experimental, non-randomized, one-group pretest-posttest design with a double pretest and a 3-month follow-up in approximately 40 participants with mTBI (~20 civilians and ~20 service members). Study objectives are to explore the feasibility and early efficacy of BEST to improve psychological health outcomes in civilian and Service Member (SM) participants with mTBI who have alexithymia (poor emotional self-awareness) and emotion dysregulation. We anticipate BEST will have good feasibility and acceptability in both civilian and service member participants, and post-treatment assessments will show significant improvements in alexithymia, emotion regulation, resiliency, and affective symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Mild TBI (determined by Ohio State University TBI Identification Method)
* ≥18 years old
* U.S. resident (exclusion for California residents)
* ≥6 months post-TBI
* elevated alexithymia and emotion dysregulation (defined by >.5 standard deviation above means on the TAS-20 and DERS)
* capacity to consent
* proficient English
* if on medications that influence affect, must be stable for at least 6 weeks
* access to a device capable of video conferencing and high speed internet.

Exclusion Criteria:

* Premorbid neurological disorder other than TBI (e.g., stroke), active or uncontrolled major psychiatric disorder and/ or disorder that would pose a safety concern (e.g., borderline personality disorder)
* degenerative neurologic condition
* visual, hearing, communication, or cognitive impairments that would impede participation
* unstable or anticipated medication changes that will influence mood/ affect during study participation
* active involvement in an intensive rehabilitation program
* individuals who recently started psychotherapy (e.g., < 3 months ago)
* participant behaviors that cause concern for their ability to participate in accordance with the study requirements and protocol (e.g., unreliable correspondences, no-shows, no-replies to multiple contacts, habitual rescheduling, unable to complete study requirements in timely manner)
* concurrent participation in any other clinical trial that aims to improve mood/ behavioral functioning will be an exclusion criterion.
* participants will be excluded if at any point, they participated in TREAT (in-person clinical trial of BEST - NCT03414463)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-03-13 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Change in Toronto Alexithymia Scale-20 (TAS-20) | Baseline, Week 6, Week 12, Week 24
  This is a 20-item self report questionnaire comprised of three sub-constructs (Difficulty Identifying feelings, Difficulty Describing feelings, Externally-oriented Thinking). The full scale range is 20-100 (higher scores indicate higher (worse) alexithymia). Subscales are summed to compute a total score.

SECONDARY OUTCOMES:
Change in Levels of Emotional Awareness Scale (LEAS) | Baseline, Week 6, Week 12, Week 24
  Objective, performance-based measure of emotional awareness and labeling. Short hypothetical scenarios are presented and participants are asked to describe how they and others would feel in the context of the scenarios. More discrete emotions earn more points (e.g., "sad" scores better than "bad"). Participants' responses are scored with an electronic system, removing human bias and interpretation. The LEAS has parallel forms (A and B), which will alternate at testing sessions.
Change in Difficulty with Emotion Regulation Scale (DERS) | Baseline, Week 6, Week 12, Week 24
  Using a 5-point Likert scale, participants rate the frequency they utilize self-regulation behaviors in response to general emotional distress. There are 6 subscales: Lack of Emotional Awareness; Lack of Emotional Clarity; Difficulties Controlling Impulsive Behaviors when Distressed; Difficulties Engaging in Goal-Directed Behavior when Distressed; Non-acceptance of Negative Emotional Responses; and Limited Access to Effective Emotion Regulation Strategies. Items are summed to provide a Total Emotion Dysregulation score. Scores range from 5 (low) to 180 (high). Higher scores are indicative of more emotion dysregulation problems. The DERS has high internal consistency, test-retest reliability, and good construct validity.

OTHER OUTCOMES:
Change in Brief Resilience Scale (BRS) | Baseline, Week 6, Week 12, Week 24
  The BRS is a self-administered questionnaire with 6 items using a 5-point Likert-style scale to assess the ability to bounce back or recover from stress. Scores range from 6-30. Higher scores are indicative of greater resilience. Total score is determined by calculating the average across all 6 responses. Scores can then be classified as Low, Normal, or High Resilience.
Change in Positive and Negative Affect Schedule (PANAS) | Baseline, Week 6, Week 12, Week 24
  The PANAS is a 20-item subjective assessment of mood (10 items for Positive Affect [PA] and 10 for Negative Affect [NA]). Using a 5-point scale, participants rate the extent to which they have experienced each mood state during a specified time frame. Subscale scores for positive and negative affect are calculated with scores ranging from 10-50. For the Positive subscale, higher score equal more positive affect. For the negative affect subscale, higher scores are indicative of more negative affect.
Change in Patient Health Questionnaire-9 (PHQ-9) | Baseline, Week 6, Week 12, Week 24
  This self-report depression assessment uses a 3-point Likert scale (score range 0-27) with higher scores indicating greater depression severity. Participants rate the frequency of specified problems during the past 2 weeks.
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Anxiety | Baseline, Week 6, Week 12, Week 24
  The PROMIS Anxiety item bank (8a) is 8 items. The instrument measures self-reported fear (fearfulness, panic), anxious misery (worry, dread), hyperarousal (tension, nervousness, restlessness), and somatic symptoms related to arousal (racing heart, dizziness). It uses a 5-point Likert scale, ranging from never to always. Anxiety scores range from 5-40 with higher scores indicating greater severity of anxiety.
Change in Patient Reported Outcomes Measurement Information System (PROMIS) Anger | Baseline, Week 6, Week 12, Week 24
  The PROMIS Anger item bank (5a) includes 5 items. The Anger instrument assesses self-reported angry mood (irritability, frustration), negative social cognitions (interpersonal sensitivity, envy, disagreeableness), and efforts to control anger. It uses a 5-point Likert scale, ranging from never to always. Anger scores range from 5-25 with higher scores indicating greater severity of anger.
Change in Post-traumatic Stress Checklist- 5 (PCL-5) | Baseline, Week 6, Week 12, Week 24
  The PCL-5 is a 20-item, self-rating scale that provides a quick and accurate measure of PTSD symptoms. Each item corresponds to current diagnostic criteria of PTSD, and each symptom is rated in terms of frequency and severity. Scores range from 0-80 with higher scores indicating greater symptom severity.
Patient Global Impression of Change (PGIC) | Week 12 and Week 24
  The PGIC captures the patient perspective regarding the achievement of clinically important change with a single item asking perception of change across a Likert scale ranging from 1 (no change) to 7 (a great deal better and a considerable improvement).
Post-treatment Satisfaction Survey | Week 12
  Overall satisfaction and satisfaction with remote delivery will be evaluated with a 9-point scale. Participants will respond to the following statements: 1) Overall, how satisfied were you with BEST? (Overall treatment satisfaction); and 2) How satisfied were you with receiving this type of treatment remotely/ via teletherapy? (Teletherapy satisfaction). Scores on each scale range from 1-9. Lower scores indicate lower satisfaction. Higher scores indicate higher satisfaction.
Change in Neurobehavioral Symptom Inventory (NSI) | Baseline, Week 12, Week 24
  The NSI is a validated 22-item self-report measure that assesses the degree of disturbance in 3 neurobehavioral symptom domains in the past 2 weeks: somatic/ sensory (e.g. dizziness, balance, nausea, vision), affective (e.g., anxiety, depression, irritability, fatigue, sleep) and cognitive (e.g., concentration, forgetfulness, decision-making, slowed thinking). On this measure, respondents rate the degree of symptom severity on a five-point scale that ranges from zero (none; symptom is rarely ever present/not a problem at all) to four (very severe; symptom is almost always present/impairs performance at work, school, or home/individual probably cannot function without help). Scores range from 0 to 110, with higher scores indicative of more severe neurobehavioral symptoms.
Change in Phenotypes and exposures (PhenX) Mental Health Core Items: Alcohol Use and Substance Use | Baseline, Week 12, Week 24
  Participants will be asked their use, over the last 30 days, of alcohol (quantity and frequency) and substances (frequency).
Change in Alcohol Use Disorders Identification Test (AUDIT-C) | Baseline, Week 12, Week 24
  The AUDIT-C is a 10-item validated self-report tool developed by the World Health Organization to assess alcohol consumption, drinking behaviors, and alcohol-related problems. Scores range from 0-12 with higher scores indicating greater alcohol use and problems.
Change in Drug Abuse Screen Test (DAST-10) | Baseline, Week 12, Week 24
  This is a 10-item self-report questionnaire that provides an index of drug abuse problems. Scores range from 0-10 with higher scores indicating more drug abuse.
Change in Pain Catastrophizing Scale | Baseline, Week 12, Week 24
  This 13-item scale evaluates the thoughts and feelings people have related to their pain. Participants rate the degree to which they agree with statements describing thoughts/ feelings about their pain (e.g., I worry all the time about whether the pain will end) on a scale ranging from 0 (not at all) to 4 (all the time). The total scores range from 0-52, with higher scores indicating more severe pain catastrophizing.
Change in PROMIS Pain Intensity Short Form (3a) | Baseline, Week 12, Week 24
  This is a 3 item self-assessment of worst pain and average pain intensity in the last 7 days as well as current pain. Scores range from 3-15 with higher scores indicating greater pain severity.
Change in PROMIS Pain Interference (8a short form) | Baseline, Week 12, Week 24
  This is an eight item measure of self-reported consequences of pain on relevant aspects of a person's life and may include the extent to which pain hinders engagement with social, cognitive, emotional, physical, and recreational activities. Scores range from 6-30 with higher scores indicating more pain interference.
Change in Perth Alexithymia Questionnaire (PAQ) | Baseline, Week 12, Week 24
  This questionnaire asks about how participants perceive and experience unpleasant and pleasant emotions. Participants will be presented with statements and must indicate on a 7-point scale, how much they agree or disagree that the statement is true in describing themselves. Scores range from 24-168 with five subscale scores and a total score indicating level of alexithymia.
Change in Ambivalence over Emotional Expressiveness Questionnaire (AEQ) | Baseline, Week 12, Week 24
  This is a 14-item self-report of the degree to which one feels ambivalent about expressing emotions using a 5-point Likert scale, with higher scores indicating greater ambivalence in expression. Total scores range from 14-70.
Change in Emotional Approach Coping (EAC) | Baseline, Week 12, Week 24
  The 8-item emotional approach coping scale assesses participants' understanding and processing of emotions in general. The EAC has good internal consistency and validity. Items are rated from 1 (I usually don't do this at all) to 4 (I usually do this a lot) and averaged. Total scores range from 8- 32. Higher mean scores indicate more use of emotional approach as a coping style.
Change in UPPS-P (Negative Urgency subscale only) | Baseline, Week 12, Week 24
  This measure evaluates various domains of impulsive behavior. One of these domain subscales is negative urgency, which is the only subscale that will be administered as part of this protocol. For this 4-item subscale, participants are presented with statements for which they must rate their agreement, using a 4-point Likert scale. Scores range from 4-16. Higher scores indicate more negative urgency.
Change in Process Model of Emotion Regulation Questionnaire (PMERQ) | Baseline, Week 12, Week 24
  This questionnaire evaluates engagement and disengagement strategies that people use to regulate their negative emotions at different stages of emotion regulation (situation selection, situation modification, attentional deployment, cognitive (re)appraisal, and response modulation). Participants rate the degree of their agreement with statements using a scale that ranges from -3 (Strongly Disagree) to 3 (Strongly Agree).
Change in Multidimensional Assessment of Interoceptive Awareness (MAIA) | Baseline, Week 12, Week 24
  The MAIA comprises 37 items on eight scales, conceptually organized in five dimensions: (a) Awareness of body sensations (Noticing scale), (b) emotional reaction and attentional response to sensations (Not-Distracting and Not-Worrying scales), (c) capacity to regulate attention (Attention Regulation scale), (d) awareness of mind-body integration (Emotional Awareness, Self-Regulation, and Body Listening scales), and (e) trusting body sensations (Trusting scale). Total scores range from 0-185. Higher score indicate greater interoceptive awareness.
Change in NIH Toolbox Loneliness | Baseline, Week 12, Week 24
  This 5 item measure of loneliness asks about the frequency with which participants felt different aspects of loneliness over the last month using a 5-point scale (1=Never to 5=Always). Total scores range from 5-25. Higher scores indicate more feelings of loneliness.

CONTACTS AND LOCATIONS:
Overall Officials: Flora Hammond, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States